CLINICAL TRIAL: NCT00606697
Title: Vestipitant and Vofopitant 2 Day PSG Study for Insomnia
Brief Title: A Study With GW597599 And GR205171: Potential New Drugs For The Treatment Of Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: NKI110334
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Primary Insomnia Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — vofopitant; vestipitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall study (Active Comparator): Male and female subjects, 18-64 years of age (inclusive), with a primary diagnosis of primary insomnia
  Interventions: Drug: GR205171; Drug: GW597599

INTERVENTIONS:
Drug: GR205171 — 10 milligrams (mg)
Drug: GW597599 — 15 mg

SUMMARY:
Patients with Primary Insomnia will be treated with GW597599 and GR205171 to evaluate the efficacy in the sleep difficulties associated with insomnia

ELIGIBILITY:
Inclusion Criteria:

* The subject must be able to read and understand the informed consent form and provide written informed consent, indicating the subjects understanding of the purpose of the study and willingness to comply with all study procedures described in the protocol, including all sleep-laboratory restrictions and procedures.
* Subject is a male or female outpatient, at least 18 years of age and <65 years.
* Diagnosis of primary insomnia, as defined by Diagnostic and Statistical Manual of Mental Disorders-Text Revision (DSM-IV-TR) criteria 307.42. A complaint of difficulty initiating or maintaining sleep or of non-restorative sleep, which lasts for at least 3 months preceding screening along with clinically significant distress or impairment in social, occupational, or other important areas of functioning. The disturbance in sleep does not occur exclusively during the course of another sleep disorder or occur exclusively during the course of another mental disorder. Lastly, the disturbance is not due to the direct physiological effects of a substance or a general medical condition.
* The subjects self-reported sleep history includes at least three months of a usual TST of less than 6 hours, SOL of at least 30 minutes and at least 3 awakening per night in at least 3 nights per week.
* On two screening PSGs (on single-blinded placebo administration at each night):

  * TST between 240 and 390 minutes inclusive on both nights.
  * Mean LPS of 30 minutes or more, but not < 20 minutes on either night.
  * Mean WASO of 60 minutes or more, with neither night < 45 minutes.
* Time in bed between 6.5 and 8.5 hours for at least 5 nights per week over the preceding 3 months
* Bed time between 21.00 and 24.00 hours that does not vary by more than ±2 hour preceding 3 months
* Women of childbearing potential must commit to consistent and correct use of an acceptable method of birth control; GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of a physician, are as follows:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses)
  * Child-bearing potential, has a negative serum pregnancy test result at screen and a negative urine dipstick pregnancy test at baseline (prior to study drug administration), and agrees to one of the following:
  * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
  * Oral contraceptives (either combined or progestogen only)
  * Double-barrier method of contraception consisting of spermicide with either condom or diaphragm
  * IUD with a documented failure rate of less than 1% per year
  * Complete abstinence from intercourse for two weeks before exposure to the investigational product, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of three days, equivalent to five half lives)

Exclusion Criteria:

* Any clinically significant psychiatric disorder other than primary insomnia as defined by DSM-IV-TR.

  - Subject must not have a Beck Depression Inventory (version II) [Beck, 1996] total score of 29 or greater at the Screening Visit. Patients scoring 17 to 28 must be confirmed by a qualified clinician to not have major depressive illness to be eligible.
* Symptoms/signs that are consistent with any primary sleep disorder other than primary insomnia, e.g., sleep apnea, restless leg syndrome, circadian rhythm sleep disorder.
* History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence (with the exception of tobacco use) within the past 12 months as defined by DSM-IV-TR.
* Positive urine drug screen (i.e., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, or opiates) or alcohol breath test at screening. No repeat test allowed.
* Any clinically significant unstable medical or surgical condition (treated or untreated).
* Any history of a clinically significant abnormality of the neurological system (including cognitive disorders or significant head injury) or any history of seizure (excluding febrile seizure).
* Subject has an unstable medical disorder; or a disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of GW597599 or GR205171; or interfere with the accurate assessment of safety or efficacy.
* Subjects having clinically significant abnormalities in haematology, blood chemistry, ECG, urinalysis, physical exam, vital signs, or other protocol-specified screening test which are not resolved by the baseline visit.
* Subjects with a history of clinically significant hepatic, cardiac (e.g. including myocardial infarction), renal, neurologic (e.g. including seizures), cerebrovascular, metabolic or pulmonary disease.
* Any serious medical disorder or condition that would in the Investigator's opinion, preclude the administration of study medication.
* Subjects who have any laboratory value outside the sponsor-specified ranges at the Screening Visit (See Appendix 9: Laboratory Parameters). Testing may be repeated once to see if value returns to within range, but such laboratory value must be resolved by the Screening PSG session (PSG 1/2).
* Subjects who are not euthyroid as evidenced by normal TSH. Subjects maintained on thyroid medication must be euthyroid for a period of at least six months prior to the Screening Visit, with no dose changes.
* Known seropositivity for human immunodeficiency virus (HIV).
* Chronic hepatitis B and C, as evidenced by positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody.
* Subjects who have any electrocardiogram (ECG) parameter outside of the Sponsor-specified range (See Appendix 8: ECG Parameters). The ECG maybe repeated once to see if the parameter returns to within range, but any such abnormality must be resolved by the screening PSG session (Visits 2/3).
* Apnea-hypopnea index of 10 or more/hour of sleep on screening PSG Night 1. Subjects failing this criterion on Night 1 Screening PSG should not be screened on Night 2.
* Movement arousal index of 10 or more/hour of sleep on screening PSG Night 1. Subjects failing this criterion on Night 1 Screening PSG should not be screened on Night 2.
* Body mass index of 34 or more at Screening Visit.
* Nightshift or rotating-shift work within the last 2 work weeks or during the study period.
* Planned travel across more than 2 time zones during the study or in the 2 weeks prior to screening.
* Consumption of 300 mg or more per day on average of xanthine-containing beverages (e.g., coffee, cola, tea, chocolate) over the preceding 1 month [NOTE: 12 oz soda = ~50 mg, 7 oz coffee or 2 oz espresso = ~100 mg, 7 oz tea = ~75 mg of caffeine].
* Smoking more than 1 pack of cigarettes per day (20 cigarettes) on average over the preceding 1 month, or inability to stop smoking during the study.
* Typical consumption of more than 7 (women) or 14 (men) alcoholic units in any week, or more than 2 (women) or 3 (men) alcoholic units in any single day, over the preceding 1 month [NOTE: 1 unit = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor].
* Regular intentional napping, i.e., more than 2 naps per week
* Use of any psychotropic medications or other medications, including over-the-counter (OTC) and herbal products, that may affect sleep/wake function within 2 weeks or 5 half-lives (whichever is longer) prior to screening or need to use any of these medications at any time during the study.
* Any history of depot neuroleptic use
* All other (non-psychotropic) drugs metabolised via the P450 3A4 pathway and CYP3A4 inducers/inhibitors must be discontinued from screening and are not allowed for the duration of the study. See the list in Study Reference Manual.
* Subjects (i.e. asthmatics) who have used systemic corticosteroids within 1 week or 5 half-lives (whichever is longer) prior to the screening visit.
* Participation in investigational trial involving NK1 antagonist (including GW679769) in the past or use of any investigational drug within 30 days or 5 half-lives of the study compound or participation in an investigational trial within 30 days prior to the Screening Visit.
* Subjects who have had hypersensitivity or intolerance to NK1 antagonists including GW597599 and GR205171.
* Subjects who, in the opinion of the investigator, would be noncompliant with the visit schedule or study procedures.
* Women having a positive serum HCG pregnancy test at Screening Visit, a positive urine pregnancy dipstick at randomization, or who are lactating or planning to become pregnant within the 3 months following the Screening Visit.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.
* An unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2007-12-19 (Actual); Primary Completion 2008-05-07 (Actual); Study Completion 2008-05-07 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time (TST) from PSG recording | Night 1 and Night 2 of every treatment period (Up to Day 63)
  TST was defined as the total amount of time (measured in minutes) that was actually spent sleeping the previous night as recorded daily in the participant's sleep diary. The score was derived by a central polysomnography (PSG) reader and was analyzed as the mean of the PSG TST recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used.
Latency to Persistent Sleep (LPS) from PSG recording | Night 1 and Night 2 of every treatment period (Up to Day 63)
  LPS was defined as the amount of time measured in minutes it takes to fall asleep as the point at which 10 minutes of uninterrupted sleep has begun as determined based on PSG objective assessments of sleep disturbance. PSG recording was performed. The score was derived by a central polysomnography reader and was analyzed as the mean of the PSG TST recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used.
Wake time after sleep onset (WASO1) from PSG recording | Night 1 and Night 2 of every treatment period (Up to Day 63)
  WASO was the time in minutes scored as wake between the onset of persistent sleep and lights on, where the onset of persistent sleep was the beginning of the first continuous 20 epochs (10 minute) scored as non-wake. Mean values were calculated based on 2 treatment PSG nights. The score was derived by a central polysomnography reader and was analyzed as the mean of the PSG TST recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used.

SECONDARY OUTCOMES:
PSG measures of sleep continuity: wake during sleep (WDS) | Night 1 and Night 2 of every treatment period (Up to Day 63)
  WDS was the duration, in minutes, of wakefulness from persistent sleep onset to final epoch of sleep. An awakening was defined as a PSG recording of at least one wake epoch, bracketed by an epoch of stage 1, 2, or stage 3/4 of non- REM sleep or REM sleep. The score was derived by a central PSG reader and was analyzed as the mean of the PSG WDS recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used. This data was not collected.
PSG measures of sleep continuity: wake after sleep (WAS) | Night 1 and Night 2 of every treatment period (Up to Day 63)
  WAS was defined as the duration of wakefulness (in minutes) from final epoch of sleep to lights on. The score was derived by a central PSG reader and was analyzed as the mean of the PSG recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used. This data was not collected.
PSG measures of sleep continuity: number of awakenings after sleep onset 1 | Night 1 and Night 2 of every treatment period (Up to Day 63)
  Number of times a participant awoke following sleep onset to lights on. The score was derived by a central PSG reader and was analyzed as the mean of the PSG recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used
PSG measures of sleep structure: Non-rapid eye movement (NREM) sleep time | Night 1 and Night 2 of every treatment period (Up to Day 63)
  It was defined as the duration in minutes of Non-REM sleep during time in bed (lights off to lights on). The scores were derived by a central polysomnography reader and was analyzed as the mean of the polysomnography NREM recordings obtained on two consecutive nights. If only one assessment was present for a particular polysomnography session, the score from that one assessment was used.
PSG measures of sleep structure: Slow-Wave Sleep (SWS) time (stage 3 and 4) | Night 1 and Night 2 of every treatment period (Up to Day 63)
  It was defined as the duration in minute of stage 3 or 4 duration during time in bed (lights off to lights on). The scores were derived by central polysomnography reader and was analyzed as the mean of the polysomnography, SWS recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used. The mean SWS for the nights (night 1 and night 2) was reported.
PSG measures of sleep structure: rapid eye movement (REM) sleep time | Night 1 and Night 2 of every treatment period (Up to Day 63)
  REM sleep time, also known as stage REM duration, is defined as the number of minutes of stage REM during time in bed (lights off to lights on). The scores were derived by a central PSG reader and was analyzed as the mean of the PSG, REM Activity recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used.
PSG measures of sleep structure: REM activity | Night 1 and Night 2 of every treatment period (Up to Day 63)
  REM activity was defined as the number of rapid eye movements during time in bed (from lights off to lights on). The scores were derived by a central PSG reader and was analyzed as the mean of the PSG, REM activity recordings obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used
PSG measures of sleep structure:REM density | Night 1 and Night 2 of every treatment period (Up to Day 63)
  REM density was defined as total REM activity divided by total REM time and was recorded as Number of REMA (N) per minute. The REM activity score and total REM time were derived by a central PSG reader. This ratio was calculated first for each of the relevant polysomnography reader recordings obtained on two consecutive nights, and then REM Density was analyzed as the mean of these two ratios. If it was only possible to calculate the ratio for one of the nights in a particular polysomnography session (REM activity or Total REM time was missing for one night), the ratio from that one night was used.
Post-Sleep questionnaire: TST | Day 1 and Day 2 of every treatment period (Up to Day 63)
  sTST was subjective (participant-rated) measurement of time to sleep. It was captured under the post sleep questionnaire as 'What is the total number of hours and min you slept last night?' and the response was recorded in mins. sTST was analyzed as the mean of the values obtained on two consecutive nights. If only one assessment is present for a particular PSG session, the score from that one assessment was used.
Post-Sleep questionnaire: WASO | Day 1 and Day 2 of every treatment period (upto Day 63)
  sWASO was subjective (participant-rated) measurement of number of awakening after sleep onset. It was captured under the post sleep questionnaire as 'After falling asleep for the first time, what was the total amount of time you spent awake before getting out of bed to rise for the day?' and the response was recorded in minutes. sWASO was reported as mean of the values obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used.
Post-Sleep questionnaire: Sleep Onset Latency (SOL) | Day 1 and Day 2 of every treatment period (upto Day 63)
  SOL was subjective (participant-rated) measurement of time to sleep. It was captured under the post sleep questionnaire as 'How long did it take you to fall asleep last night after the lights were turned out?' and the response was recorded in minute. SOL was analyzed as the mean of the values obtained on two consecutive nights. If only one assessment is present for a particular PSG session, the score from that one assessment was used.
Post-Sleep questionnaire: Number of awakenings | Day 1 and Day 2 of every treatment period (upto Day 63)
  Number of awakenings was subjective (participant-rated) measurement of number of awakening after sleep onset. It was captured under the post sleep questionnaire as 'Did you wake up during the night?' and How many times did you woke up during night? Number of awakenings was reported as mean of the values obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used.
Post-Sleep questionnaire: sleep quality (SQ) to be applied on each morning following PSG recording and at home during the 3-day period following each 2- night PSG sessions. | Day 1 and Day 2 of every treatment period (upto Day 63)
  Sleep quality was subjective (participant-rated) measurement. It was measured on a 0 to 10 scale, where 0 means poor and 10 means excellent. It was captured under the post sleep questionnaire as 'On a zero-to-ten scale, where zero means poor and 10 means excellent, by answering the question "please check the number that best describes the quality of your sleep". Scores were reported as mean of the values obtained on two consecutive nights. If only one assessment was present for a particular PSG session, the score from that one assessment was used
Digit Symbol Substitution Test (DSST) Score as daytime cognitive function tests on the morning following dose | Day 1 and Day 2 of every treatment period (Upto Day 63)
  The DSST test a subset of Wechsler Intelligence scale, which assesses the attention and psychomotor performance. During this test the participant needs to transcribe a geometric symbol with its corresponding Arabic number. The participant is initially shown numbers 1 to 9 and under each number there is a corresponding geometric symbol. A series of boxes with numbers on top is shown to the participant. The participants then copy the specific geometric symbol next to the number. The correct items transcribed within the time limit were used to generate the score. The range of score was 0 to 63. Higher scores were indicative of good cognitive function.
Verbal Learning Memory Test | Day 1 and Day 2 of every treatment period (upto Day 63)
  Verbal learning and memory test comprised of four subscales including total recall, delayed recall, retention score, and recognition discrimination index. The total recall score was the number of correctly reported words in each of the 3 learning trials and the score ranged from 0 to 36. The delayed recall score was the number of correctly reported words in the delayed recall test and the score ranged from 0 to 12. The retention score represented the score on the delayed recall test divided by the higher of the recall scores from learning trials 2 and 3, multiplied by 100. It was practically ranged from 0 to 100. The recognition discrimination index (RDI) was calculated by subtracting the total false positives score (semantically-related plus semantically un-related) from the total true-positives score obtained in the delayed recognition test)
Leeds Sleep Evaluation Questionnaire (LSEQ) Scale | Day 1 and Day 2 of every treatment period (upto Day 63)
  This scale evaluated the effects of the psychoactive compounds on sleep and early morning behavior. The questionnaire consisted of ten self rating; 100-mm-line analogue questions pertaining to four consecutive aspects of sleep: getting to sleep (GTS), quality of sleep (QOS), awakening from sleep (AFS) and behavior following wakefulness (BFW). Scores range between 0 and 100. Higher scores indicate better sleep and better early morning behavior. It was performed at week 8.
Mean Stanford sleepiness scale (SSS) | Day 1 and Day 2 of every treatment period (upto Day 63)
  This was a subjective scale to evaluate alertness of the participant on a 7-point scale. where 1 is "feeling active, vital, alert, wide awake", 2 is "still functioning at high levels, but not peak; able to concentrate", 3 is "awake, but relaxed; responsive but not fully alert", 4 is "somewhat foggy, let down", 5 is "foggy, losing interest in remaining awake", 6 is "sleepy, woozy, fighting sleep, prefer to lie down", and 7 is "no longer fighting sleep, sleep onset soon, having dream like thoughts". Thus the higher values were indicative of more sleepiness.
Number of participants with Adverse events and serious adverse events | Up to 6 months
  An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, or is an important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or a drug-induced liver injury.
Plasma concentration of GW597599 | (Pre-dose and 10 hour) at Night 1 and Night 2 of each visit
  Blood samples were collected, not to exceed 100 mL per participant for the study. The blood samples were collected at visit 4, 5,6,7,8 and Visit 9. PK sampling was done to measure the plasma concentration of GW597599.
Plasma concentration of GR205171 | (Pre-dose and 10 hour) at Night 1 and Night 2 of each visit
  Blood samples were collected, not to exceed 100 mL per participant for the study. The blood samples were collected at visit 4, 5,6,7,8 and Visit 9. PK sampling was done to measure the plasma concentration of GR205171.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Germany (7):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKI110334 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register